CLINICAL TRIAL: NCT02766725
Title: Development and Clinical Evaluation of Thermosensitive Gels for the Vaginal Delivery of Sildenafil Citrate on the Endometrium of Women Use Clomiphene Citrate for Induction of Ovulation
Brief Title: Thermosensitive Gels for the Vaginal Delivery of Sildenafil Citrate
Acronym: ss
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INSITU
Record Dates: First submitted 2016-05-06; First posted 2016-05-10 (Estimated); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- preparation F12 sildenafil in-situ gel group (Experimental): women received clomiphene citrate 150 mg/d in three divided doses 50 mg each starting from day 2 of menstruation for 5 days + preparation F12 sildenafil gel vaginally from day 5 to day 12 of menstrual cycle twice daily by a specific applicator (25 mg) per dose
  Interventions: Drug: preparation F12 sildenafil in situ gel
- preparation F2 sildenafil in-situ gel group (Active Comparator): women received clomiphene citrate 150 mg/d in three divided doses 50 mg each starting from day 2 of menstruation for 5 days + preparation F2 sildenafil gel vaginally from day 5 to day 12 of menstrual cycle twice daily by a specific applicator (25 mg) per dose
  Interventions: Drug: preparation F2 sildenafil in situ gel
- placebo gel group (Placebo Comparator): women received clomiphene citrate 150 mg/d in three divided doses 50 mg each starting from day 2 of menstruation for 5 days + placebo gel vaginally from day 5 to day 12 of menstrual cycle twice daily by a specific applicator
  Interventions: Drug: placebo gel

INTERVENTIONS:
Drug: preparation F12 sildenafil in situ gel — in situ vaginal gel
  Arms: preparation F12 sildenafil in-situ gel group
Drug: preparation F2 sildenafil in situ gel — in situ vaginal gel
  Arms: preparation F2 sildenafil in-situ gel group
Drug: placebo gel — vaginal gel
  Arms: placebo gel group

SUMMARY:
The aim of this study was to develop and characterize in situ thermosensitive gels for the vaginal administration of sildenafil as a potential treatment of the endometrial thinning that occurs as a result of the use of clomiphene citrate in induction of ovulation in women with World Health Organization type II EU gonadotrophic anovulation.

ELIGIBILITY:
Inclusion Criteria:

* women with polycystic ovaries

Exclusion Criteria:

* women with other causes of infertility

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The change of Doppler resistance index after the treatment | 10 days

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Soliman GM, Fetih G, Abbas AM. Thermosensitive bioadhesive gels for the vaginal delivery of sildenafil citrate: in vitro characterization and clinical evaluation in women using clomiphene citrate for induction of ovulation. Drug Dev Ind Pharm. 2017 Mar;43(3):399-408. doi: 10.1080/03639045.2016.1254239. Epub 2016 Nov 14. PMID 27783532